CLINICAL TRIAL: NCT05488964
Title: Exercised Breastmilk: A Randomised Controlled Trial on the Effect of Exercise Training During Lactation on Breastmilk Composition
Brief Title: Effect of Exercise Training on Breastmilk Composition
Acronym: MILKSHAKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 479236
Record Dates: First submitted 2022-07-06; First posted 2022-08-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Regular endurance training for 8 weeks
  Interventions: Behavioral: Exercise
- Control (No Intervention): Habitual living for 8 weeks

INTERVENTIONS:
Behavioral: Exercise — Supervised endurance training with moderate-to-high intensity 3-4 times weekly.
  Arms: Exercise

SUMMARY:
The aim of this trial is to investigate whether regular endurance exercise during the lactation period will influence breastmilk composition among individuals with overweight/obesity, and secondarily to assess if such changes impact the growth and health of the infants.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 years or older
* Body mass index ≥ 25 kg/m2 pre-pregnancy and/or BMI ≥ 28 kg/m2 postpartum
* Given birth to a singleton term (after 37 weeks + 0 days) baby
* 6-7 weeks postpartum at time of inclusion
* Exclusively breastfeeding the baby (no other foods are given) and intend to continue this practice for ≥ 8 weeks at inclusion
* Understands oral and written Norwegian

Exclusion Criteria:

* On-going pregnancy
* Known type 1 or type 2 diabetes
* Known cardiovascular disease
* High intensity exercise more than twice weekly the last three months before inclusion and/or an intention to start regular endurance training within the next 8 weeks at baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Breastmilk human milk oligosaccharide (HMO) 3'sialyllactose (3'SL) | 0 to 8 weeks
  Relative concentration of 3'SL in breastmilk

SECONDARY OUTCOMES:
Breastmilk human milk oligosaccharide (HMO) 3'sialyllactose (3'SL) | 0 to 4 weeks
  Relative concentration of 3'SL in breastmilk
Breastmilk metabolites | 0 to 8 weeks
  Relative concentrations of metabolites in breastmilk determined using untargeted metabolomics profiling (mass spectrometry)
Breastmilk metabolites | 0 to 4 weeks
  Relative concentrations of metabolites in breastmilk determined using untargeted metabolomics profiling (mass spectrometry)
Breastmilk microRNA | 0 to 8 weeks
  RNA sequencing
Breastmilk microRNA | 0 to 4 weeks
  RNA sequencing
Maternal insulin sensitivity | 0 to 8 weeks
  Homeostatic model assessment of insulin resistance (HOMA-IR)
Maternal fasting circulating insulin C-peptide concentrations | 0 to 8 weeks
  From fasting venous blood sampling
Maternal fasting circulating glucose concentrations | After 9 months from baseline
  From fasting venous blood sampling
Maternal circulating total cholesterol concentrations | 0 to 8 weeks
  From fasting venous blood sampling
Maternal circulating total cholesterol concentrations | After 9 months from baseline
  From fasting venous blood sampling
Maternal circulating high-density lipoprotein (HDL) concentrations | 0 to 8 weeks
  From fasting venous blood sampling
Maternal circulating high-density lipoprotein (HDL) concentrations | After 9 months from baseline
  From fasting venous blood sampling
Maternal circulating low-density lipoprotein (LDL) concentrations | 0 to 8 weeks
  From fasting venous blood sampling
Maternal circulating low-density lipoprotein (LDL) concentrations | After 9 months from baseline
  From fasting venous blood sampling
Maternal circulating triglycerides concentrations | 0 to 8 weeks
  From fasting venous blood sampling
Maternal circulating triglycerides concentrations | After 9 months from baseline
  From fasting venous blood sampling
Maternal glycated hemoglobin (HbA1c) | 0 to 8 weeks
  From fasting venous blood sampling
Maternal glycated hemoglobin (HbA1c) | After 9 months from baseline
  From fasting venous blood sampling
Maternal circulating high-sensitivity c-reactive protein | 0 to 8 weeks
  From fasting venous blood sampling
Maternal circulating high-sensitivity c-reactive protein | After 9 months from baseline
  From fasting venous blood sampling
Maternal total body mass | 0 to 8 weeks
  Impedance scale
Maternal total body mass | After 9 months from baseline
  Impedance scale
Maternal fat mass | 0 to 8 weeks
  Impedance scale
Maternal fat mass | After 9 months from baseline
  Impedance scale
Maternal fat-free mass | 0 to 8 weeks
  Impedance scale
Maternal fat-free mass | After 9 months from baseline
  Impedance scale
Maternal visceral fat area | 0 to 8 weeks
  Impedance scale
Maternal visceral fat area | After 9 months from baseline
  Impedance scale
Maternal bone mass | 0 to 8 weeks
  Impedance scale
Maternal bone mass | After 9 months from baseline
  Impedance scale
Maternal waist circumference | 0 to 8 weeks
  Measuring tape
Maternal waist circumference | After 9 months from baseline
  Measuring tape
Maternal cardiorespiratory fitness | 0 to 8 weeks
  Maximum oxygen uptake via direct gas exchange
Maternal cardiorespiratory fitness | After 9 months from baseline
  Maximum oxygen uptake via direct gas exchange
Maternal systolic blood pressure | 0 to 8 weeks
  Automatic cuff
Maternal systolic blood pressure | After 9 months from baseline
  Automatic cuff
Maternal diastolic blood pressure | 0 to 8 weeks
  Automatic cuff
Maternal diastolic blood pressure | After 9 months from baseline
  Automatic cuff
Maternal nutrition | 0 to 8 weeks
  Diet diary completed for four days at baseline and at study completion
Maternal physical activity | 0 to 8 weeks
  Number of steps per week, self-reported (questionnaire)
Maternal physical activity | After 9 months from baseline
  Number of steps per week, self-reported (questionnaire)
Maternal physical activity | 0 to 8 weeks
  Minutes of moderate-intensity physical activity per week, self-reported (questionnaire)
Maternal physical activity | After 9 months from baseline
  Minutes of high-intensity physical activity per week, self-reported (questionnaire)
Maternal psychological well-being | 0 to 8 weeks
  Self-reported (questionnaire)
Maternal psychological well-being | After 9 months from baseline
  Self-reported (questionnaire)
Infant total body mass | 0 to 8 weeks
  Impedance scale
Infant total body mass | After 9 months from baseline
  Impedance scale
Infant fat mass | 0 to 8 weeks
  Impedance scale
Infant fat mass | After 9 months from baseline
  Impedance scale
Infant muscle mass | 0 to 8 weeks
  Impedance scale
Infant muscle mass | After 9 months from baseline
  Impedance scale
Infant bone density | 0 to 8 weeks
  Impedance scale
Infant bone density | After 9 months from baseline
  Impedance scale
Infant hydration status | 0 to 8 weeks
  Impedance scale
Infant hydration status | After 9 months from baseline
  Impedance scale
Infant total body mass (trajectories) | Infant age 4 weeks
  From health records
Infant length (trajectories) | Infant age 4 weeks
  From health records
Infant head circumference (trajectories) | Infant age 4 weeks
  From health records
Infant total body mass (trajectories) | Infant age 6 weeks
  From health records
Infant length (trajectories) | Infant age 6 weeks
  From health records
Infant head circumference (trajectories) | Infant age 6 weeks
  From health records
Infant total body mass (trajectories) | Infant age 3 months
  From health records
Infant length (trajectories) | Infant age 3 months
  From health records
Infant head circumference (trajectories) | Infant age 3 months
  From health records
Infant total body mass (trajectories) | Infant age 6 months
  From health records
Infant length (trajectories) | Infant age 6 months
  From health records
Infant head circumference (trajectories) | Infant age 6 months
  From health records
Infant total body mass (trajectories) | Infant age 8 months
  From health records
Infant length (trajectories) | Infant age 8 months
  From health records
Infant head circumference (trajectories) | Infant age 8 months
  From health records
Infant total body mass (trajectories) | Infant age 10 months
  From health records
Infant length (trajectories) | Infant age 10 months
  From health records
Infant head circumference (trajectories) | Infant age 10 months
  From health records
Infant total body mass (trajectories) | Infant age 12 months
  From health records
Infant height (trajectories) | Infant age 12 months
  From health records
Infant head circumference (trajectories) | Infant age 12 months
  From health records
Infant total body mass (trajectories) | Infant age 24 months
  From health records
Infant height (trajectories) | Infant age 24 months
  From health records
Infant head circumference (trajectories) | Infant age 24 months
  From health records
Infant gut microbiota | 0 to 4 weeks
  Sequencing
Infant gut microbiota | 0 to 8 weeks
  Sequencing
Infant microRNA | 0 to 8 weeks
  Sequencing

OTHER OUTCOMES:
Exercise adherence | 0 to 8 weeks
  Number of sessions completed (logbook)
Exercise compliance | 0 to 8 weeks
  Heart rate during exercise (heart rate monitor)

CONTACTS AND LOCATIONS:
Overall Officials: Trine Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Dept Circulation and Medical Imaging, EXCAR Exercise Lab, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: IPD will be shared upon requests from researchers. The principal investigator (Trine Moholdt) will review requests.

REFERENCES:
- [Derived] Moholdt T, Ashby ER, Tommerdal KH, Lemoine MCC, Holm RL, Saetrom P, Iversen AC, Ravi A, Simpson MR, Giskeodegard GF. Randomised controlled trial of exercise training during lactation on breast milk composition in breastfeeding people with overweight/obesity: a study protocol for the MILKSHAKE trial. BMJ Open Sport Exerc Med. 2023 Oct 6;9(4):e001751. doi: 10.1136/bmjsem-2023-001751. eCollection 2023. PMID 37829712